CLINICAL TRIAL: NCT05961631
Title: The Use of Bio-Electrical Impedance Analysis Derived Parameters for Evaluating Fluid Accumulation in Critically Ill Patients Admitted to ICU: a Cohort Study
Brief Title: Bio-electrical Impedance Analysis Derived Parameters for Evaluating Fluid Accumulation
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Principal investigator, MD, PhD, Anesthesiologist Consultant, Indonesia University
Other Study IDs: IndonesiaUAnes045
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Critically Ill
Keywords: Bio-electrical Impedance Analysis; Fluid Accumulation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Positive Fluid Balance 500ml or more: Fluid Balance measured using Bio-electrical Impedance Analysis
  Interventions: Other: Bio-electrical Impedance Analysis
- Fluid Balance 500ml or less: Fluid Balance measured using Bio-electrical Impedance Analysis
  Interventions: Other: Bio-electrical Impedance Analysis

INTERVENTIONS:
Other: Bio-electrical Impedance Analysis — Variable measured: Fluid accumulation (FA), volume excess (VE), total body weight (TBW), extracellular water (ECW), intracellular water (ICW)

SUMMARY:
The purpose of this study is to assess fluid accumulation (FA) in the body using BIA (Bioelectrical Impedance Analysis) in critically ill patients treated in the ICU. This study is an observational cohort with an initial phase that analyzes prospective individual patient data

DETAILED DESCRIPTION:
This research will begin by identifying subjects through the collection of initial data. The identification of subjects will involve using BIA (Bioelectrical Impedance Analysis) equipment. Subsequently, the subjects will be divided into two groups based on the initial BIA test results of body fluid balance. The first group will comprise patients with a body fluid balance exceeding 500cc, while the second group will consist of patients with a body fluid balance of 500cc or less. Throughout the study, various BIA-derived parameters will be closely monitored for both groups, starting from the initial BIA test until the patients are discharged from the ICU or for a maximum of 7 days of ICU care from the time of the first test.

ELIGIBILITY:
Inclusion Criteria:

* New patients admitted to Intensive Care Unit Cipto Mangunkusumo Hospital and Indonesia University University
* Willing to be included in this research and signed the consent form

Exclusion Criteria:

* Obesity(BMI>35kg/m²) OR underweight (BMI < 18,5 kg/m²)
* Pregnant or Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients admitted to Intensive Care Unit Cipto Mangunkusumo Hospital and Indonesia University University
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Fluid accumulation (FA) | 1 week
  Each increase in volume excess is divided by the patient's initial body weight and expressed as a percentage. FA (fluid accumulation) is considered positive if the percentage value is greater than 5%. Conversely, FA is considered negative if the percentage value is less than 5%.

SECONDARY OUTCOMES:
volume excess (VE) | 1 week
  Fluid volume expansion outside the cells, based on the assessment by BIA (Bioelectrical Impedance Analysis), refers to the increase in fluid volume that occurs outside the cells of the body.
total body weight (TBW) | 1 week
  The total mass or weight quantity of a person is obtained from BIA (Bioelectrical Impedance Analysis) measurements.
extracellular water (ECW) | 1 week
  The amount of ECW (liters)
intracellular water (ICW) | 1 week
  The amount of ICW (liters)

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, M.D, Ph.D, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Finfer S, Myburgh J, Bellomo R. Intravenous fluid therapy in critically ill adults. Nat Rev Nephrol. 2018 Sep;14(9):541-557. doi: 10.1038/s41581-018-0044-0. PMID 30072710
- [Background] Sethakarun S, Bijaphala S, Kitiyakara C, Boongird S, Phanachet P, Reutrakul S, Pirojsakul K, Nongnuch A. Effect of bioelectrical impedance analysis-guided dry weight adjustment, in comparison to standard clinical-guided, on the sleep quality of chronic haemodialysis patients (BEDTIME study): a randomised controlled trial. BMC Nephrol. 2019 Sep 2;20(1):211. doi: 10.1186/s12882-019-1405-z. PMID 31474223
- [Background] Malbrain ML, Huygh J, Dabrowski W, De Waele JJ, Staelens A, Wauters J. The use of bio-electrical impedance analysis (BIA) to guide fluid management, resuscitation and deresuscitation in critically ill patients: a bench-to-bedside review. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):381-91. doi: 10.5603/AIT.2014.0061. PMID 25432557
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Gomez JM, Heitmann BL, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, Schols AM, Pichard C; Composition of the ESPEN Working Group. Bioelectrical impedance analysis--part I: review of principles and methods. Clin Nutr. 2004 Oct;23(5):1226-43. doi: 10.1016/j.clnu.2004.06.004. PMID 15380917
- [Background] Sanchez M, Jimenez-Lendinez M, Cidoncha M, Asensio MJ, Herrerot E, Collado A, Santacruz M. Comparison of fluid compartments and fluid responsiveness in septic and non-septic patients. Anaesth Intensive Care. 2011 Nov;39(6):1022-9. doi: 10.1177/0310057X1103900607. PMID 22165353
- [Background] Lankadeva YR, Kosaka J, Iguchi N, Evans RG, Booth LC, Bellomo R, May CN. Effects of Fluid Bolus Therapy on Renal Perfusion, Oxygenation, and Function in Early Experimental Septic Kidney Injury. Crit Care Med. 2019 Jan;47(1):e36-e43. doi: 10.1097/CCM.0000000000003507. PMID 30394921
- [Background] Nunes TS, Ladeira RT, Bafi AT, de Azevedo LC, Machado FR, Freitas FG. Duration of hemodynamic effects of crystalloids in patients with circulatory shock after initial resuscitation. Ann Intensive Care. 2014 Aug 1;4:25. doi: 10.1186/s13613-014-0025-9. eCollection 2014. PMID 25593742
- [Background] Wang N, Jiang L, Zhu B, Wen Y, Xi XM; Beijing Acute Kidney Injury Trial (BAKIT) Workgroup. Fluid balance and mortality in critically ill patients with acute kidney injury: a multicenter prospective epidemiological study. Crit Care. 2015 Oct 23;19:371. doi: 10.1186/s13054-015-1085-4. PMID 26494153
- [Background] Messmer AS, Zingg C, Muller M, Gerber JL, Schefold JC, Pfortmueller CA. Fluid Overload and Mortality in Adult Critical Care Patients-A Systematic Review and Meta-Analysis of Observational Studies. Crit Care Med. 2020 Dec;48(12):1862-1870. doi: 10.1097/CCM.0000000000004617. PMID 33009098
- [Background] Bouchard J, Soroko SB, Chertow GM, Himmelfarb J, Ikizler TA, Paganini EP, Mehta RL; Program to Improve Care in Acute Renal Disease (PICARD) Study Group. Fluid accumulation, survival and recovery of kidney function in critically ill patients with acute kidney injury. Kidney Int. 2009 Aug;76(4):422-7. doi: 10.1038/ki.2009.159. Epub 2009 May 13. PMID 19436332